CLINICAL TRIAL: NCT04935736
Title: Postoperative Pain Evaluation After Definitive Root Canal Obturation With Zinc Oxide/Eugenol-type Sealer Containing or Not 1% Prednisolone Acetate - Steroid Anti-inflammatory Agent: a Comparative, Randomized Clinical Trial.
Brief Title: Postoperative Pain After Root Canal Obturation With Sealer Containing Prednisolone.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ACTEON Group (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CORT-SP; 2021-A00525-36 (Other: French National Agency oh Health (ANSM))
Record Dates: First submitted 2021-06-09; First posted 2021-06-23 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Root Canal Obturation
Keywords: endodontic treatment; root canal sealer

STUDY DESIGN:
Intervention Model Description: Study subject (tooth) will be randomized in a 1:1 allocation ratio between the 2 treatment groups.
Who Masked: Participant
Masking Description: the participant will be blind from the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CORTISOMOL SP (Experimental): Zinc oxide/Eugenol-type sealer containing 1% Prednisolone Acetate. The sealer is used in combination with gutta percha points for the permanent obturation of root canals.
  Interventions: Device: root canal sealer : CORTISOMOL SP
- SEALITE REGULAR (Active Comparator): The Zinc oxide/Eugenol-type sealer is used in combination with gutta percha points for the permanent obturation of root canals.
  Interventions: Device: root canal sealer : SEALITE REGULAR

INTERVENTIONS:
Device: root canal sealer : CORTISOMOL SP — The participant will be treated with CORTISOMOL SP sealer in combination with gutta percha.
  Arms: CORTISOMOL SP
Device: root canal sealer : SEALITE REGULAR — The participant will be treated with SEALITE REGULAR sealer in combination with gutta percha.
  Arms: SEALITE REGULAR

SUMMARY:
The study design is a multicentric randomized controlled clinical trial. 238 subjects (teeth) requiring a primary or a secondary root canal treatment will be enrolled in 2 groups (119 in each group).

The aim is to assess the effectiveness and utility of the ancillary drug substance, prednisolone acetate (1%) contained in CORTISOMOL SP (Zinc Oxide/Eugenol-type sealer) to help to decrease the possible postoperative painful reactions after root canal treatment. SEALITE REGULAR, which has a similar formulation except it is prednisolone acetate-free, is used as the comparator sealer.

Procedures of root canal treatment will be conventional and standardized for all investigational centers. The canals will be cleaned, shaped and then obturated using a Zinc oxide/Eugenol-type sealer (CORTISOMOL SP or SEALITE REGULAR) and gutta-percha.

Patients assess their pain for 7 days after permanent root canal obturation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age > 18 years old
* Patient requiring a primary or a secondary root canal treatment on a single or multi-rooted tooth.
* Informed consent signed
* Patient with social protection.

Exclusion Criteria:

* Endodontic treatment on tooth with suspected root perforation, or immature tooth,
* Known allergy to corticosteroids, local anesthetics, or any component of the medical devices,
* Patient taking anti-pain or anti-inflammatory treatment regularly for another pathology,
* Presence of any significant medical finding or significant history such as uncontrolled systemic diseases that may impact the safety, the interpretation of the results and/or the participation of the subject in the study according to the opinion of the investigator,
* Participation in another intervnetional clinical trial or subject still within the exclusion period of a previous clinical trial,
* Vulnerable subjects referred to in articles L.1121-5 to 8 and L.1122-1-2 of the Public Health Code and article 66 of Regulation (EU) 2017/745 on medical devices are excluded from the investigation (such as known pregnancy or lactation, patients with legal protection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Post-operative pain assessed by a VAS | From the end of the root canal treatment (Day 0) to Day 7
  The pain is assessed by patients in a diary using a Visual Analogue Scale (range from 0 (= no pain) to 100 (= the worst pain)) at different times after endodontic treatment from the end of the root canal obturation to Day 7. The maximum pain felt will be compared between the 2 groups.

SECONDARY OUTCOMES:
Use of oral pain treatment | From the end of the root canal treatment (Day 0) to Day 7
  Patients reported the consumption of analgesic treatment in a diary. The proportion of patients who took oral pain medication will be compared between the 2 groups.
Number of adverse events | From the end of the root canal treatment (Day 0) to the end of follow-up visit (Day 14)
  Adverse events recorded from the endodontic treatment to the end of follow-up visit will be used to assess the safety of root canal sealers and endodontic procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Hugues Colombel, DDS, Principal Investigator — Cabinet dentaire (Rennes)
Locations (8):
- France (8):
  - Cabinet dentaire, Lamballe
  - Cabinet dentaire, Liffré
  - Cabinet dentaire, Plédran
  - Cabinet dentaire, Pluguffan
  - Cabinet dentaire, Rennes
  - CHU Rennes - Centre de Soins Dentaires, Rennes
  - Cabinet dentaire, Saint-Brieuc
  - Cabinet dentaire, Saint-Coulomb

IPD SHARING:
Plan to Share IPD: No